CLINICAL TRIAL: NCT06540924
Title: Investigation of LBX1, TIMP2, GPR126 and CHD7 Gene Polymorphisms in Adolescent Idiopathic Scoliosis Patients
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Erkan Bilgin, Specialist medical doctor, Uludag University
Other Study IDs: 2022-14/18
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Adolescent Idiopathic Scoliosis; Single Nucleotide Polymorphisms
Keywords: Adolescent idiopathic scoliosis; genetic; single nucleotide polymorphism
MeSH Terms: interventions — Polymorphism, Single Nucleotide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected from patients and control individuals using purple-capped EDTA tubes, with 2 tubes per person (totaling 6 cc). The samples were stored at -80°C until the DNA isolation process. DNA was isolated from the collected blood samples, followed by DNA quality assessment. Subsequently, analysis was conducted using primers for the SNP (single nucleotide polymorphism) regions under study on a Real-Time Polymerase Chain Reaction (RT-PCR) device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Being diagnosed with Adolescent Idiopathic Scoliosis (AIS) between the ages of 10 and 18 group. Having a Cobb angle of 10 degrees or greater on a plain radiograph. Not having any known genetic disorders. Not having any diseases known to play a role in the etiology of scoliosis (degenerative, neuromuscular, congenital scoliosis, etc., are excluded).
  Interventions: Other: single nucleotide polymorphisms
- Control group: Healthy individuals between the ages of 10-18 who do not have scoliosis by physical examination and/or imaging.
  Interventions: Other: single nucleotide polymorphisms

INTERVENTIONS:
Other: single nucleotide polymorphisms — The LBX1 (Ladybird Homeobox 1), TIMP2 (Tissue Inhibitor of Metalloprotease 2), GPR126 (G Protein-Coupled Receptor 126) and CHD7 (Chromodomain Helicase DNA Binding Protein 7) gene polymorphisms in adolescent idiopathic scoliosis patients and the control group were analyzed using real-time PCR with TaqMan probe SNP (single nucleotide polymorphism) primers (rs625039, rs11598564, rs6570507, rs121434341, rs11190870, rs8179090).

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a common disease of the spine observed in individuals aged 10-18 who typically do not have any other health issues. Despite numerous genetic studies conducted across different ethnic groups worldwide, the specific genes contributing to the development of scoliosis have not yet been definitively identified. Therefore, the aim of our study is to investigate whether there is an etiological relationship between AIS and the polymorphisms of the LBX1 (rs11190870, rs625039, rs11598564), TIMP2 (rs8179090), GPR126 (rs6570507), and CHD7 (rs121434341) genes in the Turkish population and to determine the relationship of these polymorphisms with gender, age, age at diagnosis and Cobb angle in these patients.

DETAILED DESCRIPTION:
This prospective genetic research was conducted Bursa Uludag University Faculty of Medicine, Department of Orthopedics and Traumatology. A total of 301 individuals were included in the study, comprising 201 patients aged 10-18 years diagnosed with AIS and Cobb angle of 10 degrees or more on direct radiography, no known genetic disorders and no diseases known to play a role in the etiology of scoliosis and 100 healthy controls aged 10-18 years without a diagnosis of scoliosis based on physical examination and/or imaging. In the study, the LBX1, TIMP2, GPR126 and CHD7 gene polymorphisms in AIS patients and the control group were analyzed using real-time PCR with TaqMan probe SNP (single nucleotide polymorphism) primers (rs625039, rs11598564, rs6570507, rs121434341, rs11190870, rs8179090). Subsequently, the SNP regions were confirmed by DNA sequence analysis. The obtained findings were statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

Study group

* Being diagnosed with Adolescent Idiopathic Scoliosis (AIS) between the ages of 10 and 18.
* Having a Cobb angle of 10 degrees or greater on a plain radiograph.
* Not having any known genetic disorders.
* Not having any diseases known to play a role in the etiology of scoliosis (degenerative, neuromuscular, congenital scoliosis, etc., are excluded).

Control group

* Healthy individuals who have not been diagnosed with scoliosis by physical examination and/or imaging.
* Being between the ages of 10-18

Exclusion Criteria:

Study group

* Those diagnosed with non-idiopathic scoliosis.
* Individuals who develop scoliosis after the age of 18.
* Individuals with scoliosis under the age of 10.
* Those diagnosed with a genetic disease.
* Those diagnosed with any disease known to play a role in the etiology of scoliosis.

Control group

* Those who have physical examination suspicion of scoliosis.
* Those with a Cobb angle of 10 degrees or more on plain radiographs.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals applying to Uludag University Orthopedics and Traumatology polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Investigation of LBX1, TIMP2, GPR126, and CHD7 Gene Polymorphisms in 201 Turkish Adolescents With Idiopathic Scoliosis | 12 months
  Despite numerous genetic studies conducted across different ethnic groups worldwide, the specific genes contributing to the development of scoliosis have not yet been definitively identified. Therefore, the aim of investigator is to investigate whether there is an etiological relationship between adolescent idiopathic scoliosis and the polymorphisms of the LBX1 (rs11190870, rs625039, rs11598564), TIMP2 (rs8179090), GPR126 (rs6570507), and CHD7 (rs121434341) genes in the Turkish population.

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Bilgin, Doctor, Principal Investigator — Uludag University
Locations (1):
- Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No